CLINICAL TRIAL: NCT01694329
Title: Impact of Introduction of PHiD-CV (Pneumococcal Nontypeable H. Influenza Protein D-conjugate Vaccine) for Nunavik Children, Quebec, Canada
Brief Title: Impact of Introduction of PHiD-CV for Nunavik Children, Quebec, Canada
Acronym: Nunavik2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: GSK114180
Record Dates: First submitted 2012-06-08; First posted 2012-09-27 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2015-10

CONDITIONS: Acute Upper Respiratory Infection; Acute Lower Respiratory Tract Infection; Otitis Media (OM); Invasive Pneumococcal Disease, Protection Against
Keywords: Streptococcus pneumoniae; Pneumococcal Conjugate Vaccines; Immunization; Otitis media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2006-2010 cohort: cohort of children born between 2006 and 2010, and living in Nunavik

SUMMARY:
The objective of this study is to document the residual burden of acute upper respiratory infections (AURIs), acute lower respiratory infections (ALRIs), otitis media (OMs) and auditory functional and anatomical abnormalities in children under the age of 5 years in Nunavik who will be exposed to PHiD-CV in combination with PCV-7 or PCV-13. The comparison groups will be the cohorts of children who received no PCV vaccine (those born in 1994-1996) and those exposed to PCV-7 exclusively (those born in 2003-2007).

DETAILED DESCRIPTION:
Around 1420 children born between 2006 and 2010 had been eligible to routine immunization program with pneumococcal vaccines.

The objective of this study is to document the residual burden of acute upper respiratory infections (AURIs), acute lower respiratory infections (ALRIs), otitis media (OMs) and auditory functional and anatomical abnormalities in children under the age of 5 years in Nunavik who will be exposed to PHiD-CV in combination with PCV-7 or PCV-13. The comparison groups will be the cohorts of children who received no PCV vaccine (those born in 1994-1996) and those exposed to PCV-7 exclusively (those born in 2003-2007).

The specific objectives are to measure in children under the age of 5 years in Nunavik and born in the period 2009 to 2010:

1. the incidence of invasive pneumococcal disease(IPD), AURIs, ALRIs and OMs;
2. the frequency of antibiotic treatments due to these diseases;
3. the frequency of hospitalizations and transfers to the South on account of ALRIs;
4. the frequency of tympanotomies and ventilation tube insertions;
5. the prevalence of anatomical and functional lesions of the middle ear at the age of 5 years (the main issue).

The main research hypothesis is that the incidence of AURIs, ALRIs and OMs and the prevalence of sequelae from OM decreased after the implementation of PHiD-CV in 2009, as compared with previous cohorts of children who were not exposed to this new vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Born between 2006 and 2010
* Resident in Nunavik (province of Quebec, Canada)

Exclusion Criteria:

• Not applicable

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children of Nunavik born between 2006 and 2010, who have been exposed to PHiD-CV in combination with PCV-7 or PCV-13
Sampling Method: Probability Sample
Enrollment: 1420 (Actual)
Dates: Start 2012-09; Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anatomical and functional lesions of the middle ear at the age of 5 years. | at age of 5 years old

SECONDARY OUTCOMES:
Incidence of IPDs | at age of 5 years old
Frequency of antibiotic treatments due to diseases of interest | at age of 5 years old
Frequency of hospitalizations and transfers to the South on account of ALRIs | at age of 5 years old
Frequency of tympanotomies and ventilation tube insertions | at age of 5 years old
Incidence of AURIs | at age of 5 years old
Incidence of ALRIs | at age of 5 years old
Incidence of OMs | at age of 5 years old

CONTACTS AND LOCATIONS:
Overall Officials: Philippe De Wals, MD PhD, Principal Investigator — Centre de recherche du CHUQ
Locations (1):
- Centre de recherche du CHUQ, Québec, Quebec, Canada

REFERENCES:
- [Derived] De Wals P, Zhou Z, LeMeur JB, Proulx JF. Burden of respiratory infections and otitis media in the Inuit population of Nunavik, Quebec, Canada. Int J Circumpolar Health. 2020 Dec;79(1):1799688. doi: 10.1080/22423982.2020.1799688. PMID 32730119
- [Derived] De Wals P, Lemeur JB, Ayukawa H, Proulx JF. Middle ear abnormalities at age 5 years in relation with early onset otitis media and number of episodes, in the Inuit population of Nunavik, Quebec, Canada. Int J Circumpolar Health. 2019 Dec;78(1):1599269. doi: 10.1080/22423982.2019.1599269. PMID 30924406
- [Derived] Le Meur JB, Ayukawa H, Proulx JF, De Wals P. Prevalence of middle ear abnormalities from otitis media in relation with pneumococcal vaccine use in the Inuit population of Nunavik, province of Quebec, Canada. Vaccine. 2018 Aug 16;36(34):5180-5186. doi: 10.1016/j.vaccine.2018.07.008. Epub 2018 Jul 17. PMID 30026032